CLINICAL TRIAL: NCT00016406
Title: A Comparative Randomized Study of Standard Doxorubicin and Cyclophosphamide Followed by Weekly Paclitaxel Vs. Weekly Doxorubicin and Daily Oral Cyclophosphamide Plus G-CSF Followed by Weekly Paclitaxel As Neoadjuvant Therapy For Inflammatory and Locally Advanced Breast Cancer
Brief Title: S0012 Doxorubicin, Cyclophosphamide, and Paclitaxel With or Without Filgrastim in Treating Women With Inflammatory or Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068630; S0012 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclophosphamide; Doxorubicin; Paclitaxel; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AC followed by P (Active Comparator): doxorubicin and cyclophosphamide followed by paclitaxel followed by surgery
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin; Drug: paclitaxel; Procedure: surgery
- AC+G followed by P (Experimental): weekly doxorubicin and daily cyclophosphamide with filgrastim followed by paclitaxel followed by surgery
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: doxorubicin; Drug: paclitaxel; Procedure: surgery

INTERVENTIONS:
Biological: filgrastim
  Other Names: G-CSF
  Arms: AC+G followed by P
Drug: cyclophosphamide
  Other Names: cytoxan
Drug: doxorubicin
  Other Names: Adriamycin
Drug: paclitaxel
Procedure: surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether combination chemotherapy is more effective with or without filgrastim in treating breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of combining doxorubicin, cyclophosphamide, and paclitaxel with or without filgrastim in treating women who have inflammatory or locally advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the microscopic pathologic response rates in women with inflammatory or locally advanced breast cancer treated with standard neoadjuvant doxorubicin and cyclophosphamide followed by weekly paclitaxel vs weekly doxorubicin and daily oral cyclophosphamide with filgrastim (G-CSF) followed by weekly paclitaxel.
* Compare the toxic effects of these regimens in this patient population.
* Compare the delivered dose intensity of these regimens in this patient population.
* Evaluate the association between microscopic pathologic complete response and clinical complete response at the primary tumor site in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease status (inflammatory vs other). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive doxorubicin IV followed by cyclophosphamide IV on day 1. Treatment repeats every 21 days for a total of 5 courses in the absence of disease progression or unacceptable toxicity. Three weeks after completion of doxorubicin and cyclophosphamide, patients receive paclitaxel IV over 1 hour weekly on day 1 for a total of 12 weeks.
* Arm II: Patients receive doxorubicin IV on day 1, oral cyclophosphamide on days 1-7, and filgrastim (G-CSF) subcutaneously on days 2-7. Treatment repeats weekly for a total of 15 courses of doxorubicin and cyclophosphamide and 16 courses of G-CSF in the absence of disease progression or unacceptable toxicity. One week after completion of G-CSF, patients receive paclitaxel as in arm I.

Within 3-6 weeks after completion of chemotherapy, patients with stable or responsive disease undergo surgical resection of tumor and affected nodes.

After surgery, patients may receive radiotherapy or additional chemotherapy and/or hormonal therapy at the discretion of the treating physician.

Patients are followed every 6 months for 1 year and then annually for 4 years.

PROJECTED ACCRUAL: A total of 350 patients (175 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed inflammatory or locally advanced breast cancer

  * Stage IIB (T3, N0, M0), IIIA (T3, N1-2, M0 or T0-2, N2, M0), or IIIB (T4, any N, M0 or any T, N3, M0)
  * Unresectable or otherwise appropriate for neoadjuvant therapy
  * Confirmed by core needle or incisional biopsy

    * Punch biopsy allowed if invasive disease is documented
* No distant metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Not specified

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* SGOT or SGPT no greater than 2 times ULN

Renal:

* Creatinine no greater than ULN

Cardiovascular:

* No congestive heart failure or angina pectoris
* LVEF greater than lower limit of normal

Other:

* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* HIV negative
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for breast cancer

Endocrine therapy:

* No prior hormonal therapy for breast cancer

Radiotherapy:

* No prior radiotherapy for breast cancer

Surgery:

* No prior definitive surgery for breast cancer

Other:

* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2001-05; Primary Completion 2006-09 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Comparison of microscopic pathologic response rates | no sooner than 21 days after chemo
Toxicity | during chemo and at surgery
Comparison of delivered dose intensity | after chemo
Correlation of microscopic pathologic complete response with clinical complete response at the primary tumor site | no sooner than 21 days after chemo

CONTACTS AND LOCATIONS:
Overall Officials: Georgiana K. Ellis, MD, Study Chair — Seattle Cancer Care Alliance
Locations (314):
- United States (314):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Highlands Oncology Group - Springdale, Springdale, Arkansas
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Saint Rose Hospital, Hayward, California
  - Valley Memorial Hospital, Livermore, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Highland General Hospital at St. George's University School of Medicine, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Summit Medical Center, Oakland, California
  - Comprehensive Cancer Center at Desert Regional Medical Center, Palm Springs, California
  - J.C. Robinson, M.D. Regional Cancer Center, San Pablo, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - Halifax Medical Center, Daytona Beach, Florida
  - Michael & Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Cancer Research Center of Hawaii, Honolula, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - St. Francis Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Medical and Surgical Specialists, L L C, Galesburg, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Hematology Oncology Consultants Ltd., Naperville, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers, Beech Grove, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen Health System, Goshen, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Alegent Health Community Memorial Hospital, Missouri Valley, Iowa
  - Burgess Health Center, Onawa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Siouxland Hematology-Oncology Associates at June E. Nylen Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, P.A. - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, P.A. - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, P.A. - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, P.A. - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, P.A. - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, P.A. - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Stormont-Vail Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, P.A. - Wellington, Wellington, Kansas
  - Associates in Womens Health, P.A. - North Review, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Winfield, Winfield, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Baton Rouge General Regional Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - Cancer Treatment Center at Christus Schumpert St. Mary Place, Shreveport, Louisiana
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Commonwealth Hematology-Oncology P. C. - Quincy, Quincy, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County General Hospital, Big Rapids, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Mercy Medical Center, Grand Rapids, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Metropolitan Hospital, Grand Rapids, Michigan
  - Spectrum Health Hospital - Blodgett Campus, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazooaa, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, P.C., Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Ted B. Wahby Cancer Center at Mount Clemens General Hospital, Mount Clemens, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Cancer Care Center at St. Luke's Hospital, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Woodwinds Hospital, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Gape Girardeau, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine Associates of Bozeman, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Fremont Area Medical Center, Fremont, Nebraska
  - Good Samaritan Health Systems, Kearney, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Cancer Center at Midlands Community Hospital, Papillion, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Lovelace Medical Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cancer Care Center at Catskill Regional Medical Center, Harris, New York
  - St. Vincent's Comprehensive Cancer Center - Manhattan, New York, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at Pitt County Memorial Hospital, Greenville, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, P. C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Kenton Oncology, Incorporated, Kenton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Promedica Cancer Center at Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical College of Ohio Cancer Institute, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Toledo Surgical Specialists, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - United States Air Force Medical Center Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Glesham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Institute of Oncology at Vilnius University, Portland, Oregon
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Salem Hospital Regional Cancer Center, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Oncology Services of Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Seton Shivers Cancer Program at Brackenridge Hospital, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital Regional Cancer Center, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - St. Joseph Medical Center at Franciscan Health System, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Central Washington Hospital, Wenatchee, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington
  - North Star Lodge Cancer Center, Yakima, Washington
  - Washington Hematology - Oncology Specialists, Yakima, Washington
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Result] Slovak ML, Bedell V, Lew D, et al.: Screening for clonal hematopoiesis as a predictive marker for development of t-AML following adjuvant therapy for breast cancer (S0012). [Abstract] J Clin Oncol 25 (Suppl 18): A-11051, 2007.
- [Result] Ellis GK, Barlow WE, Gralow JR, Hortobagyi GN, Russell CA, Royce ME, Perez EA, Lew D, Livingston RB. Phase III comparison of standard doxorubicin and cyclophosphamide versus weekly doxorubicin and daily oral cyclophosphamide plus granulocyte colony-stimulating factor as neoadjuvant therapy for inflammatory and locally advanced breast cancer: SWOG 0012. J Clin Oncol. 2011 Mar 10;29(8):1014-21. doi: 10.1200/JCO.2009.27.6543. Epub 2011 Jan 10. PMID 21220618
- [Derived] Slovak ML, Bedell V, Lew D, Albain KS, Ellis GK, Livingston RB, Martino S, Perez EA, Hortobagyi GN, Sher D, Stock W. Screening for clonal hematopoiesis as a predictive marker for development of therapy-related myeloid neoplasia (t-MN) following neoadjuvant therapy for breast cancer: a Southwest Oncology Group study (S0012). Breast Cancer Res Treat. 2010 Jan;119(2):391-8. doi: 10.1007/s10549-009-0597-5. PMID 19851858